CLINICAL TRIAL: NCT04540250
Title: Stratification of Oral Lesions in Methotrexate-treated Rheumatoid Arthritis Patients
Brief Title: Stratification of Oral Ulcers in Rheumatoid Arthritis Patients Kept on Methotrexate
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Magdy Ahmed, Lecturer of oral medicine, Beni-Suef University
Other Study IDs: BSU 5643
Record Dates: First submitted 2020-08-18; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Methotrexate Adverse Reaction; Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group of Rheumatoid arthritis patients: RA patients receiving MTX as monotherapy were included in the study. Patients suffering from systemic disease known to cause oral manifestations; salivary gland diseases and malignancies were excluded.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — conventional intra-oral examination and questionnaire
  Other Names: intra-oral examination

SUMMARY:
This study included rheumatoid arthritis patients receiving Methotrexate as monotherapy. All eligible patients were subjected to thorough clinical examination and full history to identify oral events. Drug history, current dose and duration of MTX were recorded.

DETAILED DESCRIPTION:
The current study was conducted in the Clinics of Oral Medicine, Faculty of Dentistry and Rheumatology, Faculty of Medicine - Cairo University from 2017 to 2019. This study followed the principles of the Helsinki Declaration and was approved by the Research ethics committee of Faculty of Dentistry, Cairo University.

RA patients receiving MTX as monotherapy were included in the study. Patients suffering from systemic disease known to cause oral manifestations; salivary gland diseases and malignancies were excluded.

All eligible patients were subjected to thorough clinical examination for the whole oral cavity. Medical history and history of any oral manifestation were recorded. Drug history, dose, and duration of MTX were recorded.

Categorical data was presented as frequencies and percentages. Continuous data was described as means and standard deviations. Means were compared by one-way ANNOVA and Student-t-test. The significance level was set at P ≤0.05. Statistical analysis was performed with IBM® SPSS® Statistics Version 25 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* patients with Rheumatoid arthritis using methotrexate as sole treatment

Exclusion Criteria:

* patients with Rheumatoid arthritis using any other treatments for Rheumatoid arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RA patients receiving MTX as monotherapy were included in the study. Patients suffering from systemic disease known to cause oral manifestations; salivary gland diseases and malignancies were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 804 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
occurrence of oral mucositis | throughout the study time (one year)
  Clinical examination (intra-oral) and history of oral mucositis where recorded

IPD SHARING:
Plan to Share IPD: Yes